CLINICAL TRIAL: NCT06858085
Title: The Turkish Version of the Late Life Function and Disability Instrument in Geriatric Individuals With Gonarthrosis: A Validity and Reliability Study
Brief Title: The Turkish Version of the Late Life Function and Disability Instrument
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Principal Investigator, Okan University
Other Study IDs: 014
Record Dates: First submitted 2025-02-22; First posted 2025-03-05 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Disability Physical
Keywords: disability; validity; reliability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Turkish Version of the Late Life Function and Disability Instrument — The Late Life Function and Disability Instrument (LLFDI) was developed to assess significant changes in functional and disability categories

SUMMARY:
The aim of this study is to investigate the Turkish validity and reliability of the Late Life Function and Disability Instrument (LLFDI) and to provide a measurement tool for researchers who wish to work in this field within the Turkish literature.

DETAILED DESCRIPTION:
Short Physical Performance Battery (SPPB), Timed Up and Go Test (TUG), Functional Independence Measure (FIM), and Barthel Index of Activities of Daily Living (MBI), among others. However, these tests were designed without a clear theoretical or conceptual framework, and their utility and applicability are limited by the physical and cognitive condition of the individuals being assessed. There is a need for practical, adequate, tolerable, and reliable tests that provide consistent results and allow for a comprehensive evaluation of functional status and the effects of treatment.

Considering the existing tests, the Late Life Function and Disability Instrument (LLFDI) was developed by professors in the Department of Physical Therapy at Boston University to assess meaningful changes in both function and disability categories. The LLFDI has been translated into Hebrew, Swedish, French, Korean, Spanish, Canadian Portuguese, and Brazilian Portuguese, with its reliability and validity confirmed. This instrument is widely used in many countries worldwide.

However, there is currently no study on the Turkish version, validity, and reliability of the Late Life Function and Disability Instrument (LLFDI).

The aim of this study is to investigate the validity and reliability of the Turkish version of the Late Life Function and Disability Instrument (LLFDI) and to provide a measurement tool for researchers in this field to be used in the Turkish literature.

ELIGIBILITY:
Inclusion Criteria:

* over 65 years old,
* being willing and volunteer to participate in the study,
* having reading and writing skills,
* being able to read and write in Turkish,
* having a diagnosis of gonarthrosis, and
* scoring above 20 points on the Mini-Mental Test.

Exclusion Criteria:

* Having a neurological problem

Ages: 65 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of individuals aged 65 and older who have been diagnosed with gonarthrosis. Participants must be able to read and write in Turkish, have no neurological problems, and score above 20 points on the Mini-Mental Test. Only volunteers who meet the inclusion criteria will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-19 (Actual)

PRIMARY OUTCOMES:
Patient Assessment Form | Baseline
  The form, prepared by the researcher, consists of 18 questions aimed at obtaining information on the sociodemographic characteristics of patients. Sociodemographic characteristics include address, age, gender, height, body weight, occupation, education level, social security status, marital status, and dominant hand.
  Additionally, fall history, medical history, family history, and use of assistive devices will be recorded to obtain general health information.
Mini-Mental Test (MMT) | Baseline
  The Mini-Mental Test (MMT) is widely used in clinical practice for detecting cognitive impairments, monitoring the progression of dementia syndromes, and assessing responses to treatment. It is also used in epidemiological studies involving elderly individuals living in the community or in institutions.
  The test consists of 11 items grouped under five main sections:
  Orientation Registration memory Attention and calculation Recall Language The total score is 30 points, and it is one of the most commonly used tests for detecting dementia. It was first described by Folstein (1975) and later refined by Molloy et al. (1991). The test has been validated and found to be reliable in the Turkish population. However, since it was initially applicable only to educated elderly individuals, it was revised in 2008 by Keskinoglu et al. to ensure its validity and reliability for both educated and uneducated elderly populations.
Late Life Function and Disability Instrument | Baseline
  The Late Life Function and Disability Instrument (LLFDI) was developed to assess significant changes in functional and disability categories.
  The function component consists of 32 questions and is evaluated in three domains:
  Upper extremity function (7 questions: F1, F3, F5, F6, F13, F16, F17) Basic lower extremity function (14 questions: F2, F10, F11, F12, F14, F15, F18, F21, F22, F23, F25, F26, F28, F31) Advanced lower extremity function (11 questions: F4, F7, F8, F9, F19, F20, F24, F27, F29, F30, F32) Each question is scored using a 5-point rating scale.
  The disability component consists of 16 questions, evaluated in two dimensions:
  Frequency Limitation Both dimensions use a 5-point rating scale. The total score of the scale is 100, with higher scores indicating better functional status.
  The scale was originally developed in the United States by Jette et al. in 2002
Barthel Activities of Daily Living Index | Baseline
  The Barthel Index assesses an individual's ability to perform daily activities independently, such as:
  Eating Using the toilet Bathing Moving indoors and outdoors
  The total score is 100, and the dependency levels are classified as follows:
  0-20 points → Completely dependent 21-61 points → Severely dependent 62-90 points → Moderately dependent 91-99 points → Mildly dependent 100 points → Fully independent The Barthel Index (BI) was developed by Mahoney and Barthel in 1965. The validity and reliability of its Turkish version were studied by Küçükdeveci et al. in 2000
Functional Independence Measure | Baseline
  The Functional Independence Measure (FIM) evaluates an individual's ability to perform daily activities independently in two domains:
  Motor Cognitive
  The total score is 126, and each item is rated as follows:
  7 points → Fully independent 6 points → Modified independence 5 points → No physical assistance needed, only verbal cues 4 points → Minimal assistance (the patient performs at least 75% of the effort) 3 points → Moderate assistance (50-75% effort by the patient) 2 points → Maximum assistance (25-50% effort by the patient)
  1 point → Total assistance The scale was first developed by Karyl et al. in 1993
Lequesne Algofunctional Knee Index | Baseline
  The Lequesne Algofunctional Knee Index is designed to evaluate patients with gonarthrosis and consists of three main components:
  Pain or discomfort Maximum walking distance Activities of daily living
  The total score is 24:
  For the first and second sections, scores range from 0 (no pain or functional limitation) to 8 (severe pain or functional limitation).
  The maximum walking distance section is scored from 0 (no limitation) to 6 (walking less than 100 m).
  If the patient uses one cane or crutch, 1 point is added; if they use two canes or crutches, 2 points are added.
  Higher scores indicate worse health status. This index was developed by Lequesne et al. in 1987

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hazar Y, Atici E, Cagliyan Erdogan H, Kardes K. Cultural adaptation and Turkish version of the Late-Life Function and Disability Instrument for individuals with gonarthrosis: a validity and reliability study. Disabil Rehabil. 2025 Nov 14:1-11. doi: 10.1080/09638288.2025.2587063. Online ahead of print. PMID 41236801